CLINICAL TRIAL: NCT02010710
Title: A Multicentre Randomised Controlled Trial of an Intelligent System to Support Decision Making in the Management of Labour Using the Cardiotocogram
Brief Title: Use of Decision Support in the Management of Labour
Acronym: INFANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University of Oxford (Other); University of Birmingham (Other); University of Plymouth (Other); University of Leicester (Other); National Childbirth Trust (Unknown); K2 Medical Systems (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06/38/01
Record Dates: First submitted 2013-06-27; First posted 2013-12-13 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Fetal Intrauterine Distress First Noted During Labor and or Delivery in Liveborn Infant; Team Based on Their Existing Guidelines and the Woman Consents to Have EFM and EFM is; Possible
Keywords: continuous electronic fetal monitoring; labour; pregnancy; fetal distress
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decison support (Experimental): "Decision-support" - CTGs with the decision support software running that will alert clinicians to the presence of abnormalities in the CTG in real time.
  Interventions: Device: INFANT software
- No Decision Support (No Intervention): "No decision-support" - CTGs with no additional interpretation (UK standard care),

INTERVENTIONS:
Device: INFANT software — The decision-support software to be evaluated in INFANT has been designed to run on the K2 data collection system (Guardian®). The data collection system (Guardian®) is a system for managing information from labour monitoring. It displays the CTG on a computer screen alongside other clinical data which are collected as part of routine clinical care. As such, it replaces conventional paper labour notes, the CTG machine and other recording systems for documenting care during labour.
  Arms: Decison support

SUMMARY:
In women judged to require continuous electronic fetal heart rate monitoring (EFM) during their labour, does the addition of decision support software to aid the interpretation of the intrapartum cardiotocogram (CTG) reduce the number of 'poor neonatal outcomes'? This study is not introducing a new form of labour monitoring; it is evaluating the addition of decision-support to CTGs displayed on the Guardian™ system. Specifically comparing: "No decision-support" - CTGs with no additional interpretation (UK standard care), compared with: "Decision-support" - CTGs with the decision support software running that will alert clinicians to the presence of abnormalities in the CTG in real time. How the labour is managed is entirely up to the recruiting unit and the woman; however the allocation of decision-support or no decision-support is determined randomly by the Guardian™ system.

ELIGIBILITY:
Inclusion Criteria:

* Require continuous electronical fetal monitoring during labour

  * they have a singleton or twin pregnancy
  * they are ≥ 35 weeks' gestation (≥ 245 days)
  * there is no known gross fetal abnormality, including any known fetal heart arrhythmia such as heart block
  * they are 16 years of age or older
  * they are able to give consent to participate in the trial as judged by the attending clinicians.

Exclusion Criteria:

* • triplets or higher order pregnancy

  * criteria for EFM not met, including elective caesarean section prior to the onset of labour

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47062 (Actual)
Dates: Start 2010-01-06 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Admissions to higher level of care | within 48 hours and for longer than 48 hours
  A composite of 'poor perinatal outcome' to include (a) all deaths (intrapartum stillbirths plus neonatal deaths i.e. deaths up to 28 days after birth) except deaths due to congenital anomalies, (b) significant morbidity: neonatal encephalopathy (moderate and severe); (c) admissions to the neonatal unit within 48 hours of birth for ≥ 48 hrs with evidence of feeding difficulties, respiratory illness or encephalopathy.

SECONDARY OUTCOMES:
Neuro Development | 2 years
  PARCA-R composite score at the age of two years

OTHER OUTCOMES:
Infant outcomes | during admission and at 2 years
  * Metabolic acidosis defined as a cord-artery pH <7.05 (this is 2 standard deviations below the mean) with base deficit ≥ 12 mmol/l (this is a threshold above which the risks of neurological damage increase)
  * The distribution of cord-blood gas data for cord-artery pH
  * Apgar score <4 at 5 minutes
  * Intrapartum stillbirth
  * Neonatal death
  * Seizures
  * Resuscitation interventions
  * Admissions to neonatal unit within 48 hours of birth for at least 48 hours
  * Admissions to neonatal unit within 48 hours of birth for at least 48 hours with evidence of:
    * Encephalopathy
    * Feeding difficulties
    * Respiratory illness
  * Admission to a higher level of care
  * In the sub-set of 7,000 surviving children without any degree of encephalopathy and agreed to be followed-up at age 2 years:
    * PARCA-R composite score
    * Cerebral palsy - (determined by asking the parents if their child has Cerebral palsy)
    * Late deaths (after the neonatal period)
    * General health issues at 2 years
Mother | during admission
  * Mode of delivery
  * Any operative intervention (caesarean section and instrumental delivery) for i. fetal distress, or ii. failure to progress, or iii. combination of fetal distress and failure to progress iv. other reason
  * Any episode of fetal blood sampling
  * Episiotomy
  * Grade of caesarean section
  * Length of first stage, length of second stage, total length of labour from trial entry

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brocklehurst, Professor, Principal Investigator — University of Birmingham
Locations (21):
- Rotunda, Dublin, Ireland
- United Kingdom (20):
  - Lancashire Women's and Newborn Centre, Burnley, Lancs
  - Birmingham Women's Hospital, Birmingham
  - Royal Bolton Hospital, Bolton
  - University Hospitals Coventry & Warwick, Coventry
  - Royal Derby Hospital, Derby
  - Princess Royal, Glasgow
  - Southern General, Glasgow
  - Liverpool Women's Hospital, Liverpool
  - Chelsea and Westminster Hospital, London
  - Homerton University Hospital, London
  - Northwick Park Hospital, London
  - St Mary's Hospital, Manchester
  - Nottingham City/Queens Medical Centre, Nottingham
  - Derriford Hospital, Plymouth
  - Queen Alexandra, Portsmouth
  - Princess Anne, Southampton
  - Stoke Mandeville Hospital, Stoke Mandeville
  - University Hospital North Staffs, Stoke-on-Trent
  - Warrington Hospital, Warrington
  - Warwick Hospital, Warwick

REFERENCES:
- See also: 2017 results — https://www.ncbi.nlm.nih.gov/pubmed/28341515
- See also: 2018 results — https://www.ncbi.nlm.nih.gov/pubmed/29437032